CLINICAL TRIAL: NCT03058211
Title: Myocardial Injury in Severe Pneumococcal Pneumonia as a Cause of Mortality From Acute Cardiovascular Events
Brief Title: Myocardial Injury and Severe Pneumococcal Pneumonia
Acronym: NEUMOCAR
Status: Terminated | Type: Observational
Why Stopped: due to COVID-19 pandemia
Sponsor: Alejandro Rodriguez Oviedo , MD (Other)
Responsible Party: Sponsor-Investigator, Alejandro Rodriguez Oviedo , MD, MD,PhD, Hospital Universitari Joan XXIII de Tarragona.
Organization: Hospital Universitari Joan XXIII de Tarragona. (Other)
Other Study IDs: PI16/00486
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Pneumonia, Pneumococcal; Myocardial Ischemia
Keywords: Pneumococcal pneumonia; Acute cardiovascular events
MeSH Terms: conditions — Pneumonia, Pneumococcal; Myocardial Ischemia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pneumococcal pneumonia: Patients with community-acquired pneumonia due to S.pneumoniae. An Echocardiography will be performed to all patients (one per day during 7 days). A Cardiac magnetic resonance (MRI) will be performed during an acute episode and at month 6 since ICU admission. In addition a blood sample will be drawn daily (one per day during 7 days) to measure myocardial injury and inflammation systemic (interleukins) biomarkers.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Cardiac Magnetic resonance
- non-pneumococcal pneumonia: Patients with community-acquired pneumonia due to S.pneumoniae. An Echocardiography will be performed to all patients (one per day during 7 days). A Cardiac magnetic resonance (MRI) will be performed during an acute episode and at month 6 since ICU admission. In addition a blood sample will be drawn daily (one per day during 7 days) to measure myocardial injury and inflammation systemic (interleukins) biomarkers.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Cardiac Magnetic resonance

INTERVENTIONS:
Diagnostic Test: Echocardiography — Standard protocols
  Other Names: Heart resonance magnetic nuclear
Diagnostic Test: Cardiac Magnetic resonance — MRI with late gadolinium increase and T1 mapping
  Other Names: MRI

SUMMARY:
Hypothesis: The "novo" cardiovascular events (CVE)in patients with severe community-acquired pneumonia (CAP) are frequent (17%) and could be associated with both direct pneumococcal myocardial invasion, toxin delivery (pneumolysin) or different biomarkers (histones, NETs(neutrophil extracellular traps), IL (Interleukin)-1b,h-Fabp (heart-Fatty acid bindding protein) ).The CVE frequency and its impact on outcome in patients without prior heart disease (CP) has not been studied.

Objectives:1) To determine the incidence of myocardian injury (MI) and CVE in patients with CAP without CP evaluated by non-invasive techniques (Echocardiograph and MRI) and biomarkers levels (Tn-I (Troponin I), h-Fabp, NT-proBNP (N-terminal pro-brain natriuretic peptide) histones, NETs, IL 1b); 2) To assess if DMA and CVE are related to the etiology and their impact on outcome , 3) To investigate the presence of myocardial scarring by MRI and its relationship with etiology and MI, and 4) To identify prognostic factors of DMA and CVE to determine level of risk.

DETAILED DESCRIPTION:
Area: Intensive care unit (ICU) of the participating hospitals. Patients: Forty patients with CAP without heart disease history will be included consecutively (20 patients with pneumococcal CAP and 20 patients with non-pneumococcal CAP).Ten healthy volunteers (controls) are included.

Variables: Epidemiological, clinical and hemodynamic variables are recorded. Presence of MI and CVE measured by echocardiography and by biomarkers will be evaluated during the ICU stay. Presence of scarring miocardic by MRI technique will be determined at month 6 since ICU admission.

Statistical analysis: Categorical (Fisher's exact test) and continuous variables( Wilconxon and Anova) will be used to determine differences between them. The Pearson correlation, ROC (discriminatory power) and logistic regression analysis(independent association) will be used to determine the association between variables and outcome. A p-value of 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. - Patients admitted to the ICU due to community-acquired pneumonia according to IDSA/ATS criteria
2. - No history of heart diasese
3. - Informed consent signed

Exclusion Criteria:

1. - Hospital or ventilator-associated pneumonia
2. - Health care-associated pneumonia
3. - Viral pneumonia
4. - Bacterial/viral coinfection pneumonia
5. - History of heart disease
6. - Chronic administration of statins
7. - Chronic administration of steorids (Prednisolone more 20 mg/day or equivalent)
8. - No signed informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the intensive care unit due to severe community-acquired pneumonia
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Myocardian injury (scarring) in patients with CAP without cardiac disease (CP)history at 6 months of ICU admission | at 6 months
  MRI with late gadolinium increase and t1 mapping techniques for to detect myocardial scarring
Heart dysfunction in patients with CAP without cardiac disease (CP)history in the first week of ICU admission | at day 7 of ICU admission)
  Echocardiography with standard and strain techniques for to detect the presence of decrease in ejection fraction of both vetricules

SECONDARY OUTCOMES:
Temporal profile of the Troponin I as a cardiac injury biomarker in patients with CAP without cardiac disease (CP)history in the first week of ICU admission | once per day ( days 1 to 7 of ICU admission)
  Determination of serum troponin-I according to standard technique
Temporal profile of the N-terminal pro-brain natriuretic peptide(NT-proBNP) as a cardiac injury biomarker in patients with CAP without cardiac disease (CP)history in the first week of ICU admission | once per day (days 1 to 7 of ICU admission)
  Determination of serum N-terminal pro-brain natriuretic peptide(NT-proBNP) according to standard technique
Temporal profile of the heart- fatty acid binding protein (h-Fabp) as a cardiac injury biomarker in patients with CAP without cardiac disease (CP)history in the first week of ICU admission | once per day (days 1 to 7 of ICU admission)
  Determination of serum heart- fatty acid binding protein (h-Fabp)according to standard technique

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro H Rodriguez Oviedo, Principal Investigator — Hospital Universitari de Tarragona Joan XXIII
Locations (1):
- Critical Care Department - Hospital Universitario de Tarragona Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corrales-Medina VF, Musher DM, Shachkina S, Chirinos JA. Acute pneumonia and the cardiovascular system. Lancet. 2013 Feb 9;381(9865):496-505. doi: 10.1016/S0140-6736(12)61266-5. Epub 2013 Jan 16. PMID 23332146
- [Background] Alhamdi Y, Neill DR, Abrams ST, Malak HA, Yahya R, Barrett-Jolley R, Wang G, Kadioglu A, Toh CH. Circulating Pneumolysin Is a Potent Inducer of Cardiac Injury during Pneumococcal Infection. PLoS Pathog. 2015 May 14;11(5):e1004836. doi: 10.1371/journal.ppat.1004836. eCollection 2015 May. PMID 25973949
- [Background] Brown AO, Mann B, Gao G, Hankins JS, Humann J, Giardina J, Faverio P, Restrepo MI, Halade GV, Mortensen EM, Lindsey ML, Hanes M, Happel KI, Nelson S, Bagby GJ, Lorent JA, Cardinal P, Granados R, Esteban A, LeSaux CJ, Tuomanen EI, Orihuela CJ. Streptococcus pneumoniae translocates into the myocardium and forms unique microlesions that disrupt cardiac function. PLoS Pathog. 2014 Sep 18;10(9):e1004383. doi: 10.1371/journal.ppat.1004383. eCollection 2014 Sep. PMID 25232870
- [Background] Lee YJ, Lee H, Park JS, Kim SJ, Cho YJ, Yoon HI, Lee JH, Lee CT, Park JS. Cardiac troponin I as a prognostic factor in critically ill pneumonia patients in the absence of acute coronary syndrome. J Crit Care. 2015 Apr;30(2):390-4. doi: 10.1016/j.jcrc.2014.12.001. Epub 2014 Dec 4. PMID 25534985
- Available data/document: Study Protocol: PI16/00486 — http://www.iispv.cat — Protocol in Spanish language
- Available data/document: Informed Consent Form: PI16/00486 — http://www.iispv.cat — Informed consent form in Spanish language